CLINICAL TRIAL: NCT01871311
Title: A Phase I Study of the BCR-ABL Tyrosine Kinase Inhibitor Nilontinib and Cetuximab in Patients With Solid Tumors That Can be Treated With Cetuximab
Brief Title: A Phase I Study of Nilontinib and Cetuximab in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary investigator left the institution.
Sponsor: Georgetown University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0039
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer; Head and Neck Cancer
Keywords: metastatic Kras wildtype; squamous cell carcinoma; cetuximab; nilotinib
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — nilotinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib + Cetuximab (Experimental): All patients with receive Nilotinib BID for a 28-day cycle + Cetuximab 400 mg/m2 on day 1 dose then 250 mg/m2 weekly
  Interventions: Drug: Nilotinib + Cetuximab

INTERVENTIONS:
Drug: Nilotinib + Cetuximab — Nilotinib BID for a 28-day cycle + Cetuximab 400 mg/m2 on day 1 dose then 250 mg/m2 weekly
  Three dose levels for nilotinib:
  Dose level -1 200-mg daily Dose level 1 200-mg BID Dose level 2 300-mg BID
  Cycle duration will be 4 weeks, with weekly evaluation of toxicity. Assessment of tumor progression will occur every 2 cycles. Subjects will be treated until disease progression or cessation due to intolerable toxicity.

SUMMARY:
The purpose of this study is to determine the recommended Phase II dose of nilotinib when used in combination with cetuximab in the treatment of patients with recurrent and/or metastatic Kras wildtype colorectal cancer or squamous cell carcinoma of the head and neck.

DETAILED DESCRIPTION:
ABL1 has been suggested to play a key role in the resistance mechanism to anti EGFR therapy in cancer. Therefore, this study aims to evaluate the safety and possible effect of targeting both EGFR using cetuximab along with ABL1 using nilotinib. Correlative studies assess the changes in tumor proteome in response to therapy and magnitude of ADCC as a marker of antibody activity.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent and/or metastatic Kras wildtype colorectal cancer or squamous cell carcinoma of the head and neck
2. Previous therapy:

   1. Patients must have progressed after standard therapy for metastatic/recurrent disease, including irinotecan and oxaliplatin-containing regimens for patients with CRC and platinum-containing regimens for patients with H&NSCC.
   2. Patients may have received cetuximab or panitumumab previously
3. Ability to swallow medication tablets by mouth (which may include taking nilotinib mixed in apple sauce)
4. At least one measurable lesion by RECIST criteria
5. A tumor lesion that can be readily biopsied using a core needle via clinical exam or image-guidance.
6. Over the age of 18 years and able to provide informed consent
7. Adequate kidney, liver, and bone marrow function as follows:

   1. Hemoglobin >/= 8.0 gm/dL
   2. Absolute neutrophil count >/= 1500
   3. Platelet count >/= 100,000
   4. Creatinine within institutional normal limits or glomerular filtration rate > 60
   5. Total bilirubin f. AST and ALT
8. Life expectancy of greater than 3 months
9. ECOG performance status
10. Normal left ventricular ejection fraction, defined as EF > 50%

Exclusion Criteria:

1. Chemotherapy or surgery within 4 weeks prior to treatment start
2. Radiation treatment within 3 weeks prior to treatment start
3. Prior therapy with nilotinib, ponatinib, dasatinib, or imatinib
4. Untreated brain metastases or neurologically unstable central nervous system metastases; CNS metastases will be considered stable if there is no new nor enlarging lesions for one month, and the patient remains off steroids and anti-epileptics for the same time period
5. Any severe or uncontrolled medical condition or other condition that could affect participation in this study, including: unstable angina, uncontrolled hypertension, serious uncontrolled cardiac arrhythmia, uncontrolled infection, or myocardial infarction
6. Diarrhea > Grade 1 at baseline
7. Concomitant medication or herbal therapy known to inhibit CYP3A4
8. Gastrointestinal tract disease resulting in the inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease
9. Ongoing ventricular cardiac dysrhythmias of NCI CTCAE grade >/= 2
10. Subjects with a history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation >/= 3 beats in a row)
11. Serious cardiac arrhythmia requiring medication
12. QTc interval > 500 msec
13. Female patients who are pregnant or breast feeding, or adults who are of reproductive potential and are unwilling to refrain from conceiving a child during study treatment
14. Patients unwilling or unable to comply with the protocol, or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 18 months
  The dose at which </= 1 out of 6 subjects experiences a dose limiting toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Ann W Gramza, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No